CLINICAL TRIAL: NCT05865028
Title: Phase II A Proof of Concept Trial Investigating Safety and Efficacy of APG-157 in Oral Dysplasia
Brief Title: A Proof of Concept Trial Investigating Safety and Efficacy of APG-157 in Oral Dysplasia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Elizabeth J Franzmann (Other)
Collaborators: Aveta Biomics, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Elizabeth J Franzmann, Professor, University of Miami
Organization: University of Miami (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20221112; NCI-2023-04230 (Registry Identifier: NCI Clinical Trials Reporting Program (NCI CTRP))
Record Dates: First submitted 2023-05-09; First posted 2023-05-18 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-12

CONDITIONS: Oropharyngeal Dysplasia; Oral Cavity Dysplasia; Oral Carcinoma in Situ

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- APG-157 Therapy (Experimental): Participants will receive APG-157 for up to 12 weeks.
  Interventions: Drug: APG-157

INTERVENTIONS:
Drug: APG-157 — Participants will take 200mg (2 x 100mg pastilles) of APG-157 therapy orally (PO) three times daily during each 4-week cycle for up to three cycles. Cycle three is optional.

SUMMARY:
The purpose of this study is to assess whether APG-157 can reduce the tumor size in participants with the study disease. Another purpose is to find out about the effects of APG-157 on certain tumor markers and oral rinses in participants with the study disease.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients age > 18 years with biopsy-proven moderate to severe oral dysplasia or carcinoma in situ (CIS) and a visible lesion. Sites include all oral cavity as well as oropharyngeal dysplasia that is accessible in the outpatient clinic.
2. Histologically proven oral cavity or oropharyngeal moderate or severe dysplasia/CIS as diagnosed by standard pathological methods and a visible lesion on oral exam.
3. Measurable disease - minimum lesion size of 8 x 3 mm before initial biopsy
4. Willing to provide blood, oral rinse and tissue from diagnostic biopsies
5. Leukocytes >=3,000/microliter
6. Absolute neutrophil count >= 1,000/microliter, Platelets >= 100,000/microliter, Total bilirubin =< 1.5 x institutional upper limit of normal (ULN), aspartate aminotransferase (AST), serum glutamic-oxaloacetic transaminase (SGOT), alanine aminotransferase (ALT) and serum glutamic pyruvic transaminase (SGPT) =< 1.5 x institutional upper limit of normal (ULN). Exceptions to this Inclusion Criteria can be made if labs are deemed not clinically significant by the principal investigator (PI).
7. Willing to use adequate contraception, subject or partner has had a vasectomy or partner is using effective birth control or is post-menopausal for the duration of the study.
8. Able to take oral medication.
9. Able to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Pregnant women.
2. Subjects who have had surgery of the oral cavity, teeth, or gums within the previous 8 weeks excluding biopsies and tooth extractions.
3. Subjects who have had a fracture of the mandible or maxilla within the previous 8 weeks.
4. Inability to complete enrollment forms due to any mental status or language problems (e.g. dementia, head injury, overall illness).
5. History of prior head and neck squamous cell carcinomas (HNSCC) unless curatively treated 1 year or more prior.
6. Use of chemotherapy and/or radiation for any malignancy (excluding nonmelanoma skin cancer and cancer confined to organs with removal as only treatment) in the past 2 years.
7. Subjects with other related diseases or the oral cavity or oropharynx, as determined to be significant by the PI.
8. History of allergic reactions attributed to compounds of similar chemical composition to Curcumin (turmeric).
9. Active or chronic liver disease, evidence of hepatitis (infectious or autoimmune), cirrhosis or portal hypertension. Exceptions to this Exclusion Criteria can be made if patient status is deemed not clinically significant by the PI.
10. Severe thrombocytopenia increasing the risk of biopsy.
11. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, uncontrolled congestive heart failure, unstable angina pectoris, uncontrolled cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-05-24 (Actual); Primary Completion 2027-05-24 (Estimated); Study Completion 2028-05-24 (Estimated)

PRIMARY OUTCOMES:
Pathologic Response Rate | Up to 12 weeks
  The pathologic response rate among participants receiving study treatment will be assessed. The pathologic response rate is defined as the percentage of participants with mild or no dysplasia after receiving study therapy. Response will be assessed on the basis of clinical, radiologic, molecular and pathologic criteria consistent with Response Evaluation Criteria in Solid Tumors (RECIST) v.1.1 criteria, per physician discretion.

SECONDARY OUTCOMES:
Clinical Response Rate | Up to 12 weeks
  The clinical response rate among participants receiving study treatment will be assessed. The clinical response rate is defined as the percentage of participants with complete response (CR) and/or partial response (PR) after receiving study therapy. Response will be assessed on the basis of clinical, radiologic, molecular and pathologic criteria consistent with Response Evaluation Criteria in Solid Tumors (RECIST) v.1.1 criteria.
Change in Lesion Appearance Before and After Protocol Therapy | Baseline, 12 weeks post-intervention, Up to 28 months
  Change in lesion appearance will be assessed using criteria consistent with Response Evaluation Criteria in Solid Tumors (RECIST) v.1.1 criteria, found at time of oral exam per physician discretion.
Number of Treatment-Related Adverse Events and Serious Adverse Events | Up to 16 weeks
  The number of treatment-related adverse events (AEs) and serious adverse events (SAEs) in participants receiving protocol therapy will be assessed using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 5, per physician discretion.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth J Franzmann, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No